CLINICAL TRIAL: NCT01141088
Title: Clinical Outcomes of Endoscopic Bilateral Stent-in-stent Placement Versus Side-by-side Method With Newly Designed Metallic Stent for Malignant Hilar Biliary
Brief Title: Two Bilateral Metal Stenting in Hilar Malignancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Tae Hoon Lee, MD, PhD, Soon Chun Hyang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCH-2010-02
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Malignant Hilar Stricture; Bilateral Stent Insertion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral stent-in-stent insertion (Experimental): The passage of the bilateral metal stent across the stricture, stent-in-stent method.
  Interventions: Procedure: Bilateral stent-in-stent insertion; Procedure: Bilateral side-by-side insertion
- Bilateral side-by-side insertion (Active Comparator): The passage of the bilateral metal stent across the stricture, side-by-side method.
  Interventions: Procedure: Bilateral stent-in-stent insertion; Procedure: Bilateral side-by-side insertion

INTERVENTIONS:
Procedure: Bilateral stent-in-stent insertion — Following negotiation of both IHD by two guidewires, inserted 1st stent to left IHD side. After deployment of the 1st stent across the hilar stricture, the remaining guide wire across the 1st stent was carefully withdrawn using an ERCP catheter without pulling it back completely. Then that guidewie was inserted under fluoroscopic guidance into the undrained right IHD through the central portion of the 1st stent. The 2nd cross-wired stent was then introduced over a guidewire through the central open mesh and then was deployed into the right IHD, so that the central portion of the 2nd stent overlapped the central portion of the 1st stent, forming a Y-shape.
  Other Names: SIS
Procedure: Bilateral side-by-side insertion — Following the introduction of two guidewires, the first stent was pushed and deployed into the left hepatic duct as possible, and then subsequently the second stent was pushed and deployed into the right hepatic duct, using the same method. In tight stricture during a guidewire manipulation, pneumatic biliary balloon dilation prior to insertion of first stent was performed. All stents were positioned above the level of the papilla, with their distal ends at the same level as possible. The diameter of the stent used in each case (8 or 10 mm) depended on the maximum diameter of the common bile duct (CBD).
  Other Names: SBS

SUMMARY:
The overall median survival of nonresectable malignant hilar obstruction in most series has been less than 6 months. Most patients with malignant hilar obstruction present with advanced disease, making allative endoscopic drainage the principal therapeutic option. However, the optimal endoscopic management strategy is contentious. In malignant hilar obstruction, exclusively endoscopic placement of bilateral metal stents has been considered very difficult and complex, and it may require multiple procedures, with an increased risk of complications and mortality. To overcome this difficulty and strategize plan of management, the investigators evaluated the technical and clinical efficacy of endoscopic bilateral placement of newly designed stents, Y-configuration, followed by side-by-side insertion in failure of stent-in-stent method for the management of malignant hilar obstruction.

DETAILED DESCRIPTION:
1. Stent-in-stent (SIS) placement Following negotiation of both intrahepatic bile ducts (IHD) by two guidewires, inserted 1st stent to left IHD side. The central portion of the 1st stent was crossed over the right-side guide wire to access the contralateral ductal system across the central cross-wired portion using the right-side guide wire as a target. After deployment of the 1st stent across the hilar stricture, the remaining guide wire across the 1st stent was carefully withdrawn using an ERCP catheter without pulling it back completely. Then that guidewie was inserted under fluoroscopic guidance into the undrained right IHD through the central portion of the 1st stent. The 2nd cross-wired stent was then introduced over a guidewire through the central open mesh and then was deployed into the right IHD, so that the central portion of the 2nd stent overlapped the central portion of the 1st stent, forming a Y-shape. If selective insertion of a guide wire into the left IHD was difficult at first, the guidewire and the 1st stent were inserted into the right IHD first and then attempts were made to insert the guide wire and a stent into the left IHD. If contralateral guide wire cannulation failed after the 1st stent placement, the stricture was dilated up to 4 or 6 mm using a balloon catheter (Hurricane biliary balloon dilatation catheter; Boston Scientific) over the guide wire. Alternatively, a second intervention for contralateral stent placement was allowed 2-3 days after expansion of the 1st endoscopic stent.
2. Side-by-side (SBS) placement Bilateral SBS stent placement was performed as follows. The stricture was first negotiated by inserting a guidewire into both IHD using the same method. Following the introduction of these two guidewires, the first stent was pushed and deployed into the left hepatic duct as possible, and then subsequently the second stent was pushed and deployed into the right hepatic duct, using the same method. During the deployment of the first stent, the second stent was preloaded on a guidewire to facilitate the bilateral SBS stent placement. Endoscopic dilatation of stricture before deployment of stents has not been routinely performed in primary procedures. In tight stricture during a guidewire manipulation, pneumatic biliary balloon dilation prior to insertion of first stent was performed. All stents were positioned above the level of the papilla, with their distal ends at the same level as possible. The diameter of the stent used in each case (8 or 10 mm) depended on the maximum diameter of the common bile duct (CBD).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* patient with malignant hilar obstruction

Exclusion Criteria:

* refuse to participate in this study
* refuse to provide informed consent
* Karnofsky score < 60%
* physically unfit for endoscopic procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | within 24 hr
  Passage of the double stent across the stricture,along with flow of contrast medium and/or bile through the stent.
  Adequate expansion: 70% of maximal expanded diameter was dilated within 24 hr.

SECONDARY OUTCOMES:
Early complications | within 30 days after stent insertion
  Early complications such as pancreatitis, cholecystitis, cholangitis, jaundice, or external or internal stent migration within 30 days after stent insertion.
Late complications | after 30 days following stent insertion
  Late complications were defines as complications such as pancreatitis, cholecystitis, cholangitis, jaundice, or stent migration after 30 days following stent insertion.
Median stent patency | up to 1 year, from stent insertion to the occlusion of the stent
Median survival | 1 year, from stent insertion to the death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Moon, MD, PhD, Principal Investigator — Soon Chun Hyang University College of Medicine, Bucheon Hospital, Bucheon, South Korea
Locations (2):
- South Korea (2):
  - Soon Chun Hyang University College of Medicine, Bucheon Hospital, Bucheon-si
  - Soon Chun Hyang University College of Medicine, Cheonan Hospital, Cheonan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee TH, Moon JH, Choi JH, Lee SH, Lee YN, Paik WH, Jang DK, Cho BW, Yang JK, Hwangbo Y, Park SH. Prospective comparison of endoscopic bilateral stent-in-stent versus stent-by-stent deployment for inoperable advanced malignant hilar biliary stricture. Gastrointest Endosc. 2019 Aug;90(2):222-230. doi: 10.1016/j.gie.2019.03.011. Epub 2019 Mar 21. PMID 30905729